CLINICAL TRIAL: NCT07196761
Title: Effect of Whole-body Vibration on Postmenopausal Constipation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nouran Mohamed Sabry, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005907
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bowel care advice group (Active Comparator): The participants will receive general bowel care advice only for 6 weeks.
  Interventions: Other: Bowel care advice
- Whole body vibration and bowl care advice group (Experimental): The participants will be subjected to whole-body vibration therapy for 25-minute/session , 3 times per week for 6 weeks in addition to general bowel care advice.
  Interventions: Other: Bowel care advice; Device: Whole-body vibration

INTERVENTIONS:
Other: Bowel care advice — It includes: - Encourage adequate fiber intake (20 to 35 grams) each day.
  * Avoid caffeine - containing foods and beverages
  * Drink at least 1.5 to 2 liters of water/day
  * Proper defecation position such as, sitting with knees higher than hips (use a foot stool or other flat, stable object if necessary) , lean forward and put elbows on knees, relax and bulge out the stomach and straighten the spine
Device: Whole-body vibration — Crazy fit massager (made in China ) with platform surface size (65 cm X 35 cm ) base height 20 cm, heavy-duty motor wattage: 200 - 500 watts, will be used to provide whole body vibration for the participants in the experimental group, for 25 minutes, 3 times per week for 6 weeks.
  Arms: Whole body vibration and bowl care advice group

SUMMARY:
This study will be conducted to investigate the effect of whole-body vibration on postmenopausal constipation

DETAILED DESCRIPTION:
Constipation is common in menopause with prevalence ranging from 4% to 29% in various parts of the world. The incidence of constipation among postmenopausal women has been reported to be 37.3%. It can affect the physical, mental and social well-being of women; it reduces individual productivity and creates a significant burden on society and disrupting women's quality of life.

Postmenopausal constipation needs to be treated as it can cause serious problems as hemorrhoids, anal fissures, pelvic organ prolapse and severe pain during defecation.

Laxatives can prevent constipation but its overuse may lead to dependency and decreased bowel function . Also, it may cause some side effects as rectal bleeding, bloody stools, severe cramps or pain, weakness or unusual tiredness, unexplained changes in bowel patterns, severe diarrhea, weakness or unusual tiredness.

Whole body vibration strengthens smooth muscles through oscillation, which causes muscles to rapidly contract and relax. This has been shown to significantly improve the condition of those with chronic functional constipation.

Whole body vibration can aid in minimizing the build up of toxins because it increases blood flow and prevent accumulation of wastes in the colon. Also, it improves gut microbiota that aid in digestion due to increased intestinal permeability.

Few studies have investigated the effect of whole body vibration specifically on postmenopausal woman. So, this study will be conducted to investigate the effect of the whole body vibration on functional constipation in postmenopausal women to provide an insight for the benefits of such intervention in the management of postmenopausal constipation.

ELIGIBILITY:
Inclusion Criteria:

* Fifty postmenopausal women are clinically diagnosed as having functional constipation after menopause (at least one year after stoppage of last menstrual cycle)
* Their age will be ranged from 50 to 60 years old.
* Their body mass index will not exceed 30 kg/m2.
* They will not receive any medical treatment.
* All of them should have at least two criteria of Rome III diagnostic criteria of constipation.

Exclusion Criteria:

* Irritable bowel syndrome or anal fissures.
* Genital organ prolapse as rectocele.
* Any neurological diseases, spinal diseases or spinal deformities.
* History of bowel surgery.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Patient Assessment of Constipation Symptom (PAC - SYM) | 6 weeks
  It is a reliable and valid tool to measure the patient's perspective constipation symptoms in terms of frequency and severity. It is a 12- item that is divided into three symptom subscales: abdominal (four items); rectal (three items); and stool (five items). Items are scored on 5-point Like scales, with scores ranging from 0 to 4 (0 = 'symptom absent', 1 = 'mild', 2 = 'moderate', 3 = 'severe' and 4 = 'very severe'). A mean total score in the range of 0-4 is generated by dividing the total score by the number of questions completed; the lower the total score, the lower the symptom burden.

SECONDARY OUTCOMES:
Patient Assessment of Constipation quality of life (PAC - QOL) | 6 weeks
  The PAC-QOL questionnaire is used to evaluate the quality of life of patients having constipation. It is a brief but comprehensive tool which evaluates constipation through daily individual health assessment and functioning. This questionnaire consists of 28 self-reported items which subcategorized into 4 items on physical discomfort. 8 items on psychosocial discomfort, 5 items on treatment satisfaction, and finally 11 items on worries and discomfort. The overall score ranges from 0 -16. The higher the score, the higher the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Azza Kassab, Professor, Study Chair — Cairo University
Locations (1):
- Nouran Mohamed Sabry, Alexandria, Egypt